CLINICAL TRIAL: NCT03481322
Title: Low Sodium Cooking Study: Acceptance of a Low Sodium Diet in Patients With Heart Diseases: a Crossover Randomized Clinical Trial
Brief Title: Low Sodium Cooking Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5364/14
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Heart Disease
Keywords: sodium chloride; diet; cooking
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooked diet with controlled amount of salt (Active Comparator): Patients will receive intervention diet (cooked with controlled amount of salt)
  Interventions: Dietary Supplement: Cooked diet with controlled amount of salt
- Cooked without salt (Placebo Comparator): Patients will receive the standard diet (cooked without salt and 2 grams of salt separated will be added by the patient)
  Interventions: Dietary Supplement: Cooked diet with controlled amount of salt

INTERVENTIONS:
Dietary Supplement: Cooked diet with controlled amount of salt — Cooked diet with controlled amount of salt by nutritionist - 2 grams of salt per patient

SUMMARY:
The purpose of this study is to evaluate the acceptance of a salt restricted diet cooked with a controlled amount of salt in patients with heart disease. Verifying if there is difference in the acceptance of the standard and hyposodic diets cooked with controlled amount of salt.

DETAILED DESCRIPTION:
Patients will be randomized into two groups. Patients in group 1 will receive on the first day the standard hyposodic diet - cooked without salt, with 2g of salt (sachet) to be added by the patient at each meal (lunch and dinner). After the first day dinner, these patients will respond to the diet acceptance questionnaire. On the second day, patients in this same group will receive the hyposodic diet cooked with controlled amount of salt at lunch and dinner. The hyposodic diet cooked with controlled amount of salt is cooked with 2 grams of salt that is divided for all the preparations, according to standardized recipes. After dinner, the patients will respond again to the diet acceptance questionnaire, however referring to the diet received in this day.

Patients in group 2 will receive the same intervention, however changing the order of reception of the diets, so, on the first day they will receive the cooked hyposodic diet with controlled amount of salt and on the second day the standard hyposodic diet (salt sachet).

The questionnaire applied refers to the reasons for not accepting the diet. The same questionnaire will be applied twice for each patient, after each of the diets offered - standard hyposodic and hyposodic cooked with controlled amount of salt.

The amount of food that was ingested by the patients, for both diets, will be evaluated by weighing the food that remains in the thermal of each meal. Leftovers of the preparations should be stored properly in plastic bags, separated by patient and properly identified, to be weighed in an electronic scale and immediately discarded in an appropriate place. It will be noted how much the patient refused from each preparation, in grams. The value obtained will be subtracted from the quantity, in grams, of the same preparation offered to the patient. The result of this operation (amount in grams of the preparation accepted / ingested by the individual) will be converted into percent. To determine the weight of the sended food, a thermometer will be weighed, which will be sent on the day, according to the standard home measure used.

ELIGIBILITY:
Inclusion Criteria:

* cardiac patients hospitalized in a clinical unit with prescription of hyposodic diet

Exclusion Criteria:

* prescription of diet with restrictions or changes in consistency;
* patients who prefer to receive soup or other non-standard food in the diet;
* pacients without unable to respond to the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-07-08 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
percentage of dietary intake of each diet | 1 day
  The amount of food that was ingested by the patients for the two diets will be evaluated by weighing the remaining food in the thermal dish of each meal. The leftovers of the preparations will be weighed in an electronic scale and it will be noted how much the patient refused of each preparation, in grams. The value obtained will be subtracted from the quantity, in grams, of the same preparation offered to the patient. The result of this operation (amount in grams of the preparation accepted / ingested by the individual) will be converted into percent.

SECONDARY OUTCOMES:
difference in the acceptance of standard and hyposodic diets cooked with controlled amount of salt | 2 days
  Comparison of the percentages of acceptance of the two diets, in total weight of the day and analysis if there was difference between the preparations

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil